CLINICAL TRIAL: NCT00002527
Title: Colorectal Adenoma Chemoprevention Trial Using Aspirin: A Phase III Study
Brief Title: Aspirin in Treating Patients With Colorectal Cancer That Has Been Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CALGB-9270; CLB-9270; E-C9270; NCCTG-949251; NCI-P93-0048; CDR0000078380 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): 325 mg/day PO
  Interventions: Drug: aspirin
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: aspirin
  Arms: Aspirin
Other: placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of aspirin may be an effective way to prevent the recurrence of polyps in colorectal cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of aspirin in treating patients who have stage I, stage II, or stage III colorectal cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether aspirin administered at a dose of 325 mg/day will decrease the number and size of new adenomas in patients with Dukes' A/B1/B2/C colorectal cancer who have undergone curative surgical resection. II. Assess whether this dose of aspirin will increase disease-free survival in these patients.

OUTLINE: Randomized, double-blind study. Arm I: Chemoprevention. Enteric-coated Aspirin, ASA, NSC-27223. Arm II: Control. Placebo, PLCB.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented colorectal cancer that has been curatively resected, including: Dukes' A/B1 (T1-2, N0, M0) Dukes' B2/C (T3, N0, M0 and any T, N1, M0) disease-free more than 5 years post-resection Colonoscopy to the cecum (or small bowel anastomosis) with removal of all polyps required within 4 months of entry Preparation must be adequate to visualize mucosa and discern the presence of no further polyps No familial polyposis (more than 100 polyps at time of resection) No history of inflammatory bowel disease including ulcerative colitis or Crohn's disease

PATIENT CHARACTERISTICS: Age: 30 to under 75 Performance status: Physician's assessment of good general health required Life expectancy: At least 5 years Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No NYHA class III/IV status No history of angina No history of MI No history of stroke or TIAs No peripheral vascular disease No bleeding diathesis including hemorrhagic stroke No prophylactic aspirin for cardiovascular disease Other: No documented peptic ulcer disease within past 15 years No aspirin sensitivity including: Aspirin-induced asthma Bronchial hyper-reactivity Urticaria Angioedema No requirement for sodium warfarin or other anticoagulant No frequent (greater than 36 times/year) NSAID use within the past 5 years No recurrent arthritis or other musculoskeletal problems No narcotic or alcohol dependency (unless there has been at least a 6-month period of abstinence) No prior or concurrent malignancy within 5 years (including metastases) except nonmelanomatous skin cancer No pregnant or nursing women Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: No concurrent enrollment in a colon cancer treatment trial or other chemoprevention trial Biologic therapy: At least 6 months since immunosuppressive therapy (i.e., azathioprine, methotrexate, cyclosporine) Chemotherapy: Prior chemotherapy allowed for patients with Dukes' B2/C colorectal cancer No concurrent chemotherapy Endocrine therapy: Prior non-immunosuppressive steroid treatment allowed Radiotherapy: Prior radiotherapy allowed for patients with Dukes' B2/C colorectal cancer No concurrent radiotherapy Surgery: Curative resection required

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 1993-05; Primary Completion 2003-03 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Reduction in size of tumors | Up to 4 years
Reduction in number of tumors | Up to 4 years
Disease free survival | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sandler, MD, MPH, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (42):
- United States (41):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Sandler RS, Halabi S, Baron JA, Budinger S, Paskett E, Keresztes R, Petrelli N, Pipas JM, Karp DD, Loprinzi CL, Steinbach G, Schilsky R. A randomized trial of aspirin to prevent colorectal adenomas in patients with previous colorectal cancer. N Engl J Med. 2003 Mar 6;348(10):883-90. doi: 10.1056/NEJMoa021633. PMID 12621132